CLINICAL TRIAL: NCT04597593
Title: Correlation Between Bleeding Complication and Treatment Failure of DOAC and Its Predictions Based on Cipherome's Pharmacogenomic Technology
Brief Title: Association Between Genetic Variant Scores and DOACs (DARES2)
Status: Completed | Type: Observational
Sponsor: Cipherome, Inc. (Industry)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: C02-002 BD001
Record Dates: First submitted 2020-10-02; First posted 2020-10-22 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Drug-Related Side Effects and Adverse Reactions; Iatrogenic Disorder
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Iatrogenic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study participants have a laboratory blood sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ADR Group: ISTH bleeding scale Major Bleeding
- Control Group: No ADR, No Treatment Failure
- Treatment Failure Group: Recurrent MI, Ischemic stroke, Other thromboembolic disorders

SUMMARY:
The study's objective is to evaluate the predictive accuracy of Cipherome's algorithm in predicting and preventing serious adverse drug reactions (ADRs) experienced by patients while on direct oral anti-coagulants (DOACs).

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient 18 years and older, who experienced a serious adverse drug reaction while taking a DOAC and is able to provide informed consent.

Exclusion Criteria:

* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients on rivaroxaban, apixaban, dabigatran, and edoxaban who experienced a serious adverse drug reaction and/or treatment failure and case-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
To determine the predictive accuracy of Cipherome's Drug Safety Score (DSS) in correlating with serious Adverse Drug Reactions associated with Direct Oral Anti-coagulants (DOACs) (rivaroxaban, apixaban, dabigatran, and edoxaban). | Within 1 year of DOAC therapy initiation
  The primary endpoint is to determine the accuracy of the DSS in predicting clinical outcomes of major bleeding per International Society of Thrombosis and Haemostatis (ISTH) criteria in subjects on Direct Oral Anti-coagulants (DOACs). The DSS is calculated on a scale of 0 to 1, with scores below 0.3 correlated with a higher risk of ADRs and scores above 0.7 correlated with a lower risk of ADRs. We will determine the DSS of all subjects who experienced major bleeding and compare it to the DSS of control subjects who did not experience bleeding.

SECONDARY OUTCOMES:
To evaluate the predictive accuracy of the DSS in correlating with serious ADRs compared to clinical tools (e.g., HAS BLED criteria). | Within 1 year of DOAC therapy initiation
  The secondary endpoint is to determine the accuracy of the DSS predicting clinical outcomes compared to clinical tools such as the HAS-BLED scoring system. A subject with a HAS-BLED score of > 4 points will be considered moderate-high risk of bleeding and a HAS-BLED score of 4 or less will be considered low risk. A DSS is calculated on a scale of 0 to 1, with scores below 0.3 correlated with a higher risk of ADRs and scores above 0.7 correlated with a lower risk of ADRs. Both DSS (low and high risk subjects) and HAS-BLED scores (low and high risk subjects) will be compared to actual clinical outcomes to assess the predictive accuracy of each scoring system.
To evaluate the predictive accuracy of the DSS in correlating with treatment failures while on Direct Oral Anti-coagulants (DOACs) | Within 1 year of DOAC therapy initiation
  The secondary endpoint is to determine the accuracy of the DSS in predicting treatment failures (e.g., recurrent MI, systemic embolism, or ischemic stroke) as compared to clinical outcomes while on DOACs. The DSS is calculated on a scale of 0 to 1, with preliminary studies demonstrating that scores below 0.3 correlated with a higher risk of ADRs and scores above 0.7 correlated with a lower risk of ADRs.

OTHER OUTCOMES:
To discover novel pharmacogenetic variants associated with Direct Oral Anti-coagulants (DOACs) | Within 1 year of DOAC therapy initiation
  Novel variants will be assessed using whole genome sequencing to evaluate the genetic pathways in individuals with serious ADRs and treatment failures. Through our analyses we intend to identify novel genetic variants in subjects with serious ADRs or treatment failure while on P2Y12 inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Ilyoung Oh, MD, Principal Investigator — SNUBH
Locations (1):
- SNUBH, Seongnam-si, Gyonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zareh M, Davis A, Henderson S. Reversal of warfarin-induced hemorrhage in the emergency department. West J Emerg Med. 2011 Nov;12(4):386-92. doi: 10.5811/westjem.2011.3.2051. PMID 22224125
- [Background] Kirley K, Qato DM, Kornfield R, Stafford RS, Alexander GC. National trends in oral anticoagulant use in the United States, 2007 to 2011. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):615-21. doi: 10.1161/CIRCOUTCOMES.112.967299. Epub 2012 Sep 4. PMID 22949490
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Jul 9;74(1):104-132. doi: 10.1016/j.jacc.2019.01.011. Epub 2019 Jan 28. No abstract available. PMID 30703431
- [Background] Bauer KA. Pros and cons of new oral anticoagulants. Hematology Am Soc Hematol Educ Program. 2013;2013:464-70. doi: 10.1182/asheducation-2013.1.464. PMID 24319220
- [Background] Xian Y, Xu H, O'Brien EC, Shah S, Thomas L, Pencina MJ, Fonarow GC, Olson DM, Schwamm LH, Bhatt DL, Smith EE, Hannah D, Maisch L, Lytle BL, Peterson ED, Hernandez AF. Clinical Effectiveness of Direct Oral Anticoagulants vs Warfarin in Older Patients With Atrial Fibrillation and Ischemic Stroke: Findings From the Patient-Centered Research Into Outcomes Stroke Patients Prefer and Effectiveness Research (PROSPER) Study. JAMA Neurol. 2019 Oct 1;76(10):1192-1202. doi: 10.1001/jamaneurol.2019.2099. PMID 31329212
- [Background] Kanuri SH, Kreutz RP. Pharmacogenomics of Novel Direct Oral Anticoagulants: Newly Identified Genes and Genetic Variants. J Pers Med. 2019 Jan 17;9(1):7. doi: 10.3390/jpm9010007. PMID 30658513
- [Background] Sennesael AL, Larock AS, Douxfils J, Elens L, Stillemans G, Wiesen M, Taubert M, Dogne JM, Spinewine A, Mullier F. Rivaroxaban plasma levels in patients admitted for bleeding events: insights from a prospective study. Thromb J. 2018 Nov 12;16:28. doi: 10.1186/s12959-018-0183-3. eCollection 2018. PMID 30455596
- [Background] Ing Lorenzini K, Daali Y, Fontana P, Desmeules J, Samer C. Rivaroxaban-Induced Hemorrhage Associated with ABCB1 Genetic Defect. Front Pharmacol. 2016 Dec 19;7:494. doi: 10.3389/fphar.2016.00494. eCollection 2016. PMID 28066243
- [Background] Ueshima S, Hira D, Kimura Y, Fujii R, Tomitsuka C, Yamane T, Tabuchi Y, Ozawa T, Itoh H, Ohno S, Horie M, Terada T, Katsura T. Population pharmacokinetics and pharmacogenomics of apixaban in Japanese adult patients with atrial fibrillation. Br J Clin Pharmacol. 2018 Jun;84(6):1301-1312. doi: 10.1111/bcp.13561. Epub 2018 Apr 16. PMID 29457840
- [Background] Shi J, Wang X, Nguyen JH, Bleske BE, Liang Y, Liu L, Zhu HJ. Dabigatran etexilate activation is affected by the CES1 genetic polymorphism G143E (rs71647871) and gender. Biochem Pharmacol. 2016 Nov 1;119:76-84. doi: 10.1016/j.bcp.2016.09.003. Epub 2016 Sep 8. PMID 27614009
- [Background] Dimatteo C, D'Andrea G, Vecchione G, Paoletti O, Cappucci F, Tiscia GL, Buono M, Grandone E, Testa S, Margaglione M. Pharmacogenetics of dabigatran etexilate interindividual variability. Thromb Res. 2016 Aug;144:1-5. doi: 10.1016/j.thromres.2016.05.025. Epub 2016 May 26. PMID 27261537
- [Background] Sychev DA, Levanov AN, Shelekhova TV, Bochkov PO, Denisenko NP, Ryzhikova KA, Mirzaev KB, Grishina EA, Gavrilov MA, Ramenskaya GV, Kozlov AV, Bogoslovsky T. The impact of ABCB1 (rs1045642 and rs4148738) and CES1 (rs2244613) gene polymorphisms on dabigatran equilibrium peak concentration in patients after total knee arthroplasty. Pharmgenomics Pers Med. 2018 Jul 25;11:127-137. doi: 10.2147/PGPM.S169277. eCollection 2018. PMID 30100750
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Selak V, Kerr A, Poppe K, Wu B, Harwood M, Grey C, Jackson R, Wells S. Annual Risk of Major Bleeding Among Persons Without Cardiovascular Disease Not Receiving Antiplatelet Therapy. JAMA. 2018 Jun 26;319(24):2507-2520. doi: 10.1001/jama.2018.8194. PMID 29946729